CLINICAL TRIAL: NCT04813575
Title: COVID 19 A Prospective Case Control Pathophysiological Study of Long Term Implications
Brief Title: COVID-19 Pathophysiology of Long Term Implications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Mohammed Alhajji, Doctor, King Faisal Specialist Hospital & Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2200055
Record Dates: First submitted 2021-02-08; First posted 2021-03-24 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Pulmonary Fibrosis; Organising Pneumonia; Thromboembolism
Keywords: Histology; COVID 19; Pulmonary fibrosis; organizing pneumonia; COVID 19 thromboembolism
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis; Bronchiolitis Obliterans; Thromboembolism; Organizing Pneumonia

STUDY DESIGN:
Intervention Model Description: Patients with COVID 19 will be followed prospectively, those who has evidence of pulmonary fibrosis after six weeks of illness will be offered cryobiopsy, and the patients who does not have significant fibrosis or do not warrant biopsy will be control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Experimental arm patients will have cryobiopsies for histological analysis of the ongoing pathology
  Interventions: Other: Cryo lung biopsies
- control group (No Intervention): This arm will be control group and will be observed prospectively

INTERVENTIONS:
Other: Cryo lung biopsies — Bronchoscopic lung biopsy utilizing the cryo technique
  Arms: Intervention arm

SUMMARY:
Coronavirus disease 2019 (COVID 19) is primarily a respiratory viral infection. At the time of writing this protocol, more than 25 million people have been affected globally. Of these, more than 850000 have died directly due to the disease. In the Kingdom of Saudi Arabia, there are as of now over 30000 cases and deaths from COVID 19. This has been declared as a Pandemic by WHO and has brought normal life to a standstill. There are many uncertainties regarding the pathophysiology and clinical course of this disease. It is estimated that 80 percent of those infected will not need special care. However, 1 in 5 (20%) patients will require hospitalization. Of these, typically, 5 percent will be critically ill and ventilated. Of those ventilated, 20 to 60 percent will die. However, this can vary from country to country due to various reasons. For example, in one study, 71.6% were hospitalized in the Kingdom of Saudi Arabia, and 4.6% were admitted to intensive care.

The rest of those who are hospitalized (95%), are at risk of having long term sequelae. From the SARS CoV infection data, 50 per cent had changes consistent with inflammatory lung disease at 4 weeks, and at 15 years, 4.6% (SD 6.4%) had pulmonary fibrosis. Middle East Respiratory Syndrome (MERS) had typical lower lobe fibrotic changes in more than one-third of the patients. SARS CoV2 virus shares 79.5% sequence identity with SARS CoV and 50% with MERS CoV. The SARS CoV2 may also have similarities in the inflammatory response; emerging data shows that COVID 19 patients also have new interstitial lung disease changes and thromboembolic disease. These patients may have long term physiological disability such as exertional hypoxia, breathlessness, reduction in static and dynamic lung volumes and diffusion factors.

There is currently no data available to predict who is at risk of developing long term chronic thromboembolic disease and interstitial lung disease. More importantly, there are no data available on the pathological changes of inflammatory lung disease. Pathologically classifying the disease may have a significant impact on the choice of the treatment for these patients who otherwise have the potential to be disabled lifelong. With appropriate phenotyping, appropriate risk reduction strategies and targeted therapies can be considered. Furthermore, studying biomarkers that could potentially identify those at-risk patients from very early on can provide an opportunity to start on the treatment very early on in the natural course of the disease history.

DETAILED DESCRIPTION:
COVID 19. A prospective case-control pathophysiological study of long term implications.

The rationale of the study To identify the phenotype of patients who would have long term complications from COVID 19 The investigators hypothesize that

1. Cytokine and inflammatory biomarkers and histopathology will allow phenotyping of patients with COVID 19 disease
2. That clinical, histopathological and radiological correlation may provide further information into the different phenotypes of COVID 19 patients.

Aim and Objectives of the study Primary objective: To phenotype COVID 19 patients based on biomarkers

Secondary objectives:

1. Risk factors for developing long term pulmonary complications
2. Risk factors for thromboembolic disease
3. Pathology of long term lung complications in COVID 19 Method

   1. Study design and setting This is a prospective cohort comparison study of patients with a confirmed diagnosis of COVID 19 clinically and with a positive Polymerase Chain Reaction (PCR) test or antibodies done later in the disease history.
   2. Study population All patients admitted to the hospital with confirmed COVID-19 infection will be approached for the recruitment in the study following appropriate consent
   3. Study assessments Baseline Assessment The following data will be collected at the baseline Clinical

      * Demographics - age, sex, BMI (if available)
      * Co-morbid conditions, especially known respiratory disease and heart failure.
      * Date of onset of symptoms
      * History of presentation and onset of the disease with important clinical features Physiological measurements
      * Inspired fraction of oxygen (FiO2), Oxygen saturation, heart rate, blood pressure and temperature at the time of enrolment
      * Method of ventilation (spontaneous, high flow nasal cannula, non-invasive ventilation, invasive ventilation, invasive ventilation + extra-corporeal membrane oxygenation)
      * Ventilatory pressures (if applicable) Investigations
      * Radiological changes - chest -x-ray and CT scan where available
      * Arterial blood gas - FiO2, pH, paO2, paCO2, HCO3, lactate- if not available, then a venous blood gas
      * Routine laboratory investigations - Hemoglobin, Lymphocyte count, Neutrophil Count, Urea, Creatinine, eGFR, ALT, AST, ALP, Bilirubin, CRP, Troponin, D-Dimer, Ferritin, NT-proBNP.
      * Cytokine assay - IL1b, IL6, MCP1, IL2ra, IL10, INFgamma levels

      Follow up at 6 - 8 weeks following discharge from the hospital

      Clinical
      * Signs and symptoms Physiological measurements
      * Oxygen saturation, heart rate and blood pressure
      * Six-minute walk test
      * Full lung function tests Investigations
      * Routine laboratory investigations - Hemoglobin, Lymphocyte count, Neutrophil Count, Urea, Creatinine, eGFR, ALT, AST, ALP, Bilirubin, CRP, Troponin, D-Dimer, Ferritin, NT-proBNP.
      * Cytokine assay - - IL1b, IL6, MCP1, IL2ra, IL10, INFgamma levels
      * Lung Ultrasound - if more than 3 B lines per field in two or more zones then proceed with CT scan
      * If there is more than 4% desaturation on a six-minute walk test, a volume CT scan with high-resolution reconstructions, where possible, a Dual-energy CT scan with Iodine mapping.
      * Echocardiogram
      * If the CT is normal, then a V/Q scan or SPECT scan to look at mismatch and shunt fraction estimation.
      * Arterial blood gas - FiO2, pH, paO2, paCO2, HCO3, lactate- if not feasible, then a venous blood gas

      Lung biopsy If the CT is abnormal, then proceed with Cryobiopsies following MDT discussion and agreement.

      Cryobiopsies will be needed in at least two of each radiological patterns of interstitial lung disease. Biopsy specimen will be examined for pathological changes, and also potential PCR testing will be done to identify any dormant SARS COV2 virus antigen presence. During bronchoscopy, a Broncho-alveolar lavage will also be done from an agreed site in the MDT discussion. Samples will be sent for cytology and microbiology.

      Follow up - 8- 10 weeks post-discharge Review patients with the results, explain results and start treatment as per the local physician's clinical decision.

      Repeat bloods
      * Routine laboratory investigations - Hemoglobin, Lymphocyte count, Neutrophil Count, Urea, Creatinine, eGFR, ALT, AST, ALP, Bilirubin, CRP, Troponin, D-Dimer, and Ferritin.
      * NT - pro BNP only if it was elevated in the first follow up. Follow up 12-week post-discharge Clinical
      * Symptoms and signs Investigations
      * Routine laboratory investigations - Hemoglobin, Lymphocyte count, Neutrophil Count, Urea, Creatinine, eGFR, ALT, AST, ALP, Bilirubin, CRP, Troponin, D-Dimer, and Ferritin.
      * NT - pro BNP only if it was elevated in the first follow up.
      * Full lung function test
      * Chest x-ray
      * Lung ultrasound

      Follow up 6 months post-discharge
      * Routine laboratory investigations - Hemoglobin, Lymphocyte count, Neutrophil Count, Urea, Creatinine, eGFR, ALT, AST, ALP, Bilirubin, CRP, Troponin, D-Dimer, and Ferritin.
      * NT - pro BNP only if it was elevated in the first follow up.
      * Full lung function test
      * Chest x-ray
      * Lung ultrasound
      * Volume CT scan with high-resolution reconstructions if possible Dual-energy CT scan with Iodine mapping.
      * If the patient had a V/Q scan, then repeat this with shunt fraction estimation. This will be the end of the trial follow up of the patients. Patients will have care as per the clinical need dictated by the physician.
   4. Data considerations

      Sample Size This is an exploratory study as there are no previous data in this population. The target sample size will be 60, with 30 patients as controls tested positive for COVID 19 disease at first follow up (6 to 8 weeks).

      Those patients who are initially enrolled in the study will be withdrawn if the patient wishes not to continue in the research or proven to be COVID negative.

      All patients admitted to the hospital will be approached for inclusion in the study. The investigators expect to recruit this number within 12 months, and the last patients follow up will be finished in 18 months.

      Statistical Analysis Descriptive statistics will be presented as proportions or means with standard deviations.

      To assess risk factors of developing complications, chi-square test, linear regression, and logistic regression methods will be used for continuous and categorical variables where appropriate multivariate modelling will also be used. Only variables with ≤10% missing data will be included in the multivariate analysis. Multiple imputations will be used to account for missing baseline data.

      A p-value of less than 0.05 will be considered statistically significant. All the statistical analysis will be performed by using the Statistical Package for the Social Sciences (SPSS) version 20 or above (IBM, USA) for Windows or by using other Statistical Package to perform exploratory data analysis and produce descriptive statistics. Normality will be tested using the skewness and kurtosis test; these parameters' values should be zero in an ideal normal distribution.

      Data Management Data will be collected by the chief investigator, principal investigator, trial coordinator and the trial team members. Patient data will be anonymized with trial number allocations.

      The data will be analyzed by the trial team and the trial statistician. This is an 18 month trial with subsequent data analysis and manuscript production.

      All patients will be assigned a unique identifying number. The database will be accessible only to authorized individuals. Appropriate database software will be used to develop the database and enter the data. Data on all the variables specified will be collected consistently. A data monitoring committee will meet periodically and review the data collection and management procedures for the completeness of coverage and data quality.

      Data usage for future studies/research

      The data will be stored for 5 years. The data will be transferred to a password only accessible drive with passwords for the clinical database and the coding database. This data storage process will be duplicated in case of data loss, and the data will be stored in a lockable office [Chief Investigators Office at King Faisal Specialist Hospital and Research Centre (KFSHRC)].

      All future publications will follow the standard procedure for studies /research at KFSHRC.
   5. Ethical considerations

   <!-- -->

   1. Confidentiality

      The confidentiality of personal information will be dealt with utmost care. All information collected will be protected, and patient anonymity ensured. No personal identifying information will be stored with the data. The information collected will not affect the safety or treatment of the patient. The study will be conducted according to the principles of Good Clinical Practice, the Declaration of Helsinki, and the rules and regulations of the Ethics committee of KFSHRC Riyadh.

      Moreover, confidentiality and anonymity will be strictly adhered to in the discussion and publication of the results. The autonomy of the patients will be observed.
   2. Patient Consent This is a prospective study recording patient's clinical details, laboratory investigations, and imaging. Most of the investigations are part of the routine care provided for a COVID 19 patient admitted to secondary care. The investigation that is not part of the routine care but is a part of the trail are Cytokine assays, which is a blood test, V/Q scan if indicated and lung biopsy.

The lung biopsy obtained using cyrobiopsy technique is an invasive procedure for selected patients within the trial cohort who have interstitial lung disease. This involves a risk of pneumothorax and bleeding. Patients will have appropriate consent for this procedure explaining the risk and benefits. Not all patients in the trial will have this intervention.

As data will be collected prospectively, the patient will be informed that data will be gathered from patient charts for the study. When the patient agrees, it will be recorded on the patient chart.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with COVID symptoms to hospitals.
* Patients >18 years old

Exclusion Criteria:

* Patients without capacity to consent
* Pulmonary oedema secondary to decompensated cardiac, renal or liver disease at the time of admission
* Interstitial lung disease at the time of presentation
* Known lymphangitis carcinomatosis
* Morbidly obese patients with BMI more than 40
* Patients with known pulmonary hypertension or if the clinician feels there are other reasons for pulmonary hypertension than cardiomyopathy secondary to COVID 19.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Post COVID 19 infection development of respiratory failure | 12- 18 months
  incidence of respiratory failure post COVID 19 infection

SECONDARY OUTCOMES:
Pathology of long term lung complications in COVID 19 | 12 - 18 months
  Histological features of pulmonary fibrosis in post-COVID infection
Risk factors for thromboembolic disease | 12-18 months
  Clinical features, cytokine assay and histopathological correlation will be used to identify risk factors for developing arterial and venous thrombotic disease

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed AlHajji, MD, Principal Investigator — King Faisal Specialist Hospital and research Centre
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Result] Spagnolo P, Balestro E, Aliberti S, Cocconcelli E, Biondini D, Casa GD, Sverzellati N, Maher TM. Pulmonary fibrosis secondary to COVID-19: a call to arms? Lancet Respir Med. 2020 Aug;8(8):750-752. doi: 10.1016/S2213-2600(20)30222-8. Epub 2020 May 15. No abstract available. PMID 32422177
- [Result] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Result] Claudia R, Sara T, GianLuca C etl. Complications and mortality of transbronchial lung cryobiopsy and surgical lung biopsy in interstitial lung diseases. Europpean Respiratory Journal. 2015 46: PA2031; DOI: 10.1183/13993003.congress-2015.PA2031.
- [Result] WHO Statement: Knowing the risks for COVID 19. https://www.who.int/indonesia/news/detail/08-03-2020-knowing-the-risk-for-covid-19.
- [Result] Alsofayan YM, Althunayyan SM, Khan AA, Hakawi AM, Assiri AM. Clinical characteristics of COVID-19 in Saudi Arabia: A national retrospective study. J Infect Public Health. 2020 Jul;13(7):920-925. doi: 10.1016/j.jiph.2020.05.026. Epub 2020 Jun 8. PMID 32534945